CLINICAL TRIAL: NCT02174952
Title: Efficacy of a Self-help Parenting Intervention for Parents of Children With ADHD in Adjunct to Pharmacotherapy
Brief Title: Self-help in Adjunct to Pharmacotherapy
Acronym: SHIP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Nottingham (Other)
Collaborators: Institute of Mental Health Nottingham (Other); National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 12031
Record Dates: First submitted 2014-06-23; First posted 2014-06-26 (Estimated); Last update posted 2014-06-26 (Estimated); Status verified 2014-06

CONDITIONS: Attention Deficit Hyperactivity Disorder (ADHD)
Keywords: Parenting interventions; ADHD; Family functioning; Parent Training
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- TAU+SH (Experimental): Families allocated to receive their usual treatment + self-help (TAU+SH) will receive 12 weeks of a self-help version of the New Forest Parenting Programme in addition to the usual treatment they are receiving from their clinician. They will also receive an introductory DVD aimed at highlighting key components of the intervention.
  Interventions: Behavioral: Self-help version of the New Forest Parenting Programme
- TAU (No Intervention): Families in the Treatment as Usual (TAU) condition will receive nothing additional to the treatment offered by their paediatrician or Child & Adolescent Mental Health Services (CAMHS) during the trial phase. Families in the TAU condition will be offered the self-help manual at the end of the trial.

INTERVENTIONS:
Behavioral: Self-help version of the New Forest Parenting Programme
  Arms: TAU+SH

SUMMARY:
Therapist-led parenting interventions have been shown to reduce symptoms of attention deficit hyperactivity disorder (ADHD) and are recommended as a first line treatment for school age children with ADHD. However, parenting interventions can be costly and impractical for parents due to factors such as time constraints and travelling costs. A self-help parent training manual has been developed and initial results have shown moderate reductions in ADHD symptoms, indicating that whilst self-help may offer a cost effective alternative to therapist led parent training interventions, it may not be sufficient to treat ADHD alone. This study therefore aims to compare the efficacy and additional benefits of the self-help intervention plus treatment as usual including pharmacotherapy with a control treatment as usual group . Families with a child aged 6-10 with a clinical diagnosis of ADHD will be recruited to the study via referrals from community paediatricians and child and adolescent mental health services. After gaining informed consent subjects will be randomised to self-help plus Treatment as usual (TAU) + or TAU (control). Those allocated to TAU+SH will be issued with the self-help manual and an introductory DVD to highlight key aspects of the intervention. Self-help intervention will last for 12 weeks. Data will be collected via standardised questionnaires completed by the parent, teacher and child and a recorded speech samples from the parent. Data will be collected at three time points; pre-intervention, post-intervention (12 weeks) and as a long term follow up (28 weeks). After completing the trial, qualitative data will be collected about participants' experience of self-help intervention.

ELIGIBILITY:
Inclusion Criteria:

* Parent/Main caregiver aged 18 years or over.
* Children aged been 6-10 years who have received a clinical diagnosis of ADHD.
* Children who are about to commence a course of medication for ADHD for the first time or a currently receiving medication for ADHD.

Exclusion Criteria:

* Parents who are not fluent in English, or unable to read English. (Due to copyright restrictions the self-help manual is only available in English.)
* Families who clinicians feel may be unable/incapable of completing the self-help intervention (e.g. where parents have severe mental illness)
* Parents who are aware that they have had previous experience of the NFPP

Ages: 6 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2012-07; Primary Completion 2014-09 (Estimated); Study Completion 2014-09 (Estimated)

PRIMARY OUTCOMES:
Efficacy subscale of the Parenting Sense of Competence Questionnaire (PSOC) | Post- Intervention (12 weeks)
  This questionnaire provides a measure of parenting confidence and satisfaction within their parenting role; parents of children with ADHD often report low parenting efficacy.

SECONDARY OUTCOMES:
Child ADHD Symptoms | 12 weeks
  Parent and teacher report according to SNAP-IV
Family Strain Index (Riley et al, 2006). | 12 weeks
Eyberg Child Behaviour Inventory (ECBI; Eyberg, 1980) | 12 weeks
Vanderbilt Diagnostic Rating Scale (Performance scale; Wolraich et al, 2003) | 12 weeks
Southampton ADHD medication behaviour and and Attitudes scale (SAMBA) | 12 weeks
Child Health and Illness Profile (parent and child report; Riley et al, 2004) | 12 weeks
Parental Expressed emotion via recorded Five Minute Speech Sample (Daley et al, 2003) | 12 weeks
General Health Questionnaire (12 item; Goldberg, 1992) | 12 weeks
Child ADHD symptoms | 28 weeks
  Parent and teacher report according to SNAP-IV
Family Strain Index (Riley et al, 2006) | 28 weeks
Eyberg Child Behaviour Inventory (ECBI; Eyberg, 1980) | 28 weeks
Vanderbilt Diagnostic Rating Scale (Performance scale; Wolraich et al, 2003) | 28 weeks
Southampton ADHD medication behaviour and and Attitudes scale (SAMBA) | 28 weeks
Child Health and Illness Profile (parent and child report; Riley et al, 2004) | 28 weeks
General Health Questionnaire (12 item; Goldberg, 1992) | 28 weeks

OTHER OUTCOMES:
Treatment Fidelity | Fortnightly throughout intervention period
  Fidelity of self-help intervention will be assessed using a parent self-report rating collected via fortnightly phone calls to parents from research/clinic staff.
Usual Treatment | Baseline, Post-intervention (12 weeks) follow-up (28 weeks)
  A treatment report form questionnaire will be used to gain information about other treatments being received for ADHD. This information will be requested initially from parents and then, with consent, from clinicians if parents feel unable/fail to provide.

REFERENCES:
- [Derived] Daley D, Tarver J, Sayal K. Efficacy of a self-help parenting intervention for parents of children with attention deficit hyperactivity disorder in adjunct to usual treatment-Small-scale randomized controlled trial. Child Care Health Dev. 2021 Mar;47(2):269-280. doi: 10.1111/cch.12825. Epub 2020 Dec 2. PMID 33159336